CLINICAL TRIAL: NCT06642909
Title: A Multicenter, Randomized, Open Label, Cyclosporine Controlled Phase II Clinical Study Evaluating the Efficacy and Safety of Zuberitamab Injection (HS006) in Patients With Primary Membranous Nephropathy
Brief Title: A Phase II Study of Zuberitamab Injection in Patients With Primary Membranous Nephropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS006-MN-01
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zuberitamab 600mg (Experimental)
  Interventions: Drug: Zuberitamab 600mg
- Zuberitamab 1000mg (Experimental)
  Interventions: Drug: Zuberitamab 1000mg
- cyclosporine (Active Comparator)
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: Zuberitamab 600mg — administered twice with a 2-week interval between each dose (i.e. D1, D15). One treatment cycle is 24 weeks
  Arms: Zuberitamab 600mg
Drug: Zuberitamab 1000mg — administered twice with a 2-week interval between each dose (i.e. D1, D15). One treatment cycle is 24 weeks
  Arms: Zuberitamab 1000mg
Drug: cyclosporine — Initial dose of 3.5 mg/kg/d, oral administration, divided into two doses, taken 12 hours apart (Q12h)
  Arms: cyclosporine

SUMMARY:
This study is a multicenter, randomized, open label, cyclosporine controlled Phase II trial aimed at evaluating the efficacy, safety, pharmacokinetics, and immunogenicity of Zuberitamab in patients with primary membranous nephropathy, and exploring the Phase III dosing regimen, sample size, and endpoint evaluation time

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and be able to complete the trial according to the protocol;
2. The age range is between 18 and 75 years old (including the critical value, subject to the day of signing the informed consent form), regardless of gender;
3. Diagnosed with primary (idiopathic) membranous nephropathy by renal biopsy before or during screening;
4. During the screening period and baseline visit, the urinary protein/creatinine ratio (UPCR) based on 24-hour urine collection should be ≥ 3.5 g/g;
5. The estimated glomerular filtration rate (eGFR) using the CKD-EPI formula is ≥ 40mL/min/1.73m2;
6. If you are taking angiotensin-converting enzyme inhibitors (ACEi) or angiotensin II receptor antagonists (ARBs), you need to maintain a stable dosage for at least 4 weeks before screening;
7. Women with fertility who have a negative pregnancy test during the screening period and before the first treatment with the investigational drug (D1 [allowed -7-day time window]) must agree to take effective contraceptive measures from the signing of the informed consent form to 6 months after the last administration; Women with fertility include all women who have had their first menstrual period and have not undergone sterilization procedures (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or have not yet reached menopause. Menopausal women are defined as having amenorrhea for at least 12 consecutive months without any other reason; Women with irregular menstrual cycles undergoing hormone replacement therapy (HRT) and serum follicle stimulating hormone (FSH) levels>35 mIU/mL; Women who are using oral, implanted, or injectable contraceptives, or using methods such as intrauterine devices, vaginal diaphragms, condoms, and spermicides for contraception, or women who have limited sexual activity and have had their sexual partners sterilized (such as vasectomy), should be considered to have fertility.

Exclusion Criteria:

1. Secondary membranous nephropathy (such as malignant tumors, systemic autoimmune diseases, drugs, etc.).
2. People with type 1 diabetes or type 2 diabetes with diabetic nephropathy (type 2 diabetics need to have renal biopsy reports within 1 year before screening).
3. Individuals with severe allergies to rituximab or other human mouse chimeric antibodies in the past (such as anaphylactic shock and angioedema) or known allergies to any ingredients or excipients of the investigational drug.
4. Individuals who have previously been resistant to cyclosporine or cyclophosphamide, or resistant to CD20 or any other therapy that leads to B cell depletion (ineffective) are identified by investigators.
5. Individuals with evidence of a >50% decrease in urine protein/creatinine ratio within the first 6 months of screening .
6. There is no evidence during the screening period to suggest that the patient is positive for PMN related antibodies.
7. Any of the following abnormal laboratory test results during screening: a. Abnormal liver function, defined as AST or ALT values>2 x upper limit of normal (ULN), or total bilirubin values>1.5 x ULN; b. Total white blood cell count<3.0 x 109/L, absolute neutrophil count<1.5 x 109/L, platelet count<75 x 109/L, or hemoglobin<90g/L.
8. Virological examination results during screening: a. Hepatitis B surface antigen (HBsAg) positive individuals; b. The patient is negative for hepatitis B surface antigen and positive for hepatitis B core antibody, and the result of further hepatitis B virus DNA test exceeds the upper limit of the hospital's reference value; c. Patients with positive hepatitis C virus (HCV) antibodies and HCV RNA; d. The human immunodeficiency virus (HIV) serum reaction is positive.
9. Suspected active or latent tuberculosis patients based on medical history or tuberculosis screening.
10. Individuals with known active bacterial, viral, fungal, mycobacterial, parasitic, or other infections (excluding fungal infections of the nail bed) or any major systemic infection requiring intravenous antibiotic treatment or hospitalization within 4 weeks prior to the baseline visit.
11. Other serious diseases that may restrict the subjects from participating in the test, such as uncontrollable diabetes; Severe heart failure (NYHA grade II or above); Acute coronary syndrome occurred within the past 6 months; Coronary revascularization such as stent implantation, coronary artery bypass surgery, and other heart and large vessel related surgeries within the past 6 months; Severe arrhythmias include frequent premature ventricular contractions, ventricular tachycardia, rapid atrial fibrillation/flutter, and severe bradycardia; Uncontrolled hypertension (greater than 150/100mmHg); Severe respiratory diseases (such as obstructive pulmonary disease and history of bronchospasm).
12. Individuals who have had or currently have malignant tumors within the past 5 years (excluding skin squamous cell carcinoma, basal cell carcinoma, and cervical carcinoma in situ that have been successfully treated and have no evidence of recurrence).
13. Those who have received live/attenuated vaccines within 4 weeks prior to the baseline visit, or those who plan to receive live vaccines during the study period;
14. Received organ/tissue transplantation or stem cell transplantation.
15. Perform any major surgical procedures within 12 weeks prior to the baseline visit or during the planned study period.
16. According to the researchers' assessment, there is a clinically significant history of drug or alcohol abuse within the 6 months prior to the baseline visit.
17. Pregnant or lactating women.
18. For those who have participated in clinical trials of other drugs and have not been screened for more than 30 days since the last administration or have 5 half lives of the original investigational drug (whichever is longer), or plan to participate in another drug clinical trial during the study period.
19. Researchers believe that there are other symptoms or conditions that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieved overall response (OR) in the urinary protein/creatinine ratio (UPCR) at week 76 | Week 76
  The proportion of subjects who achieved overall response (OR) in the urinary protein/creatinine ratio (UPCR) at week 76

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China